CLINICAL TRIAL: NCT01539759
Title: Immediate Postplacental Insertion of Intrauterine Devices at Time of Cesarean Delivery: A Randomized Clinical Trial
Brief Title: Immediate Postplacental Insertion of IUDs at Time of Cesarean Delivery: A Randomized Clinical Trial
Acronym: IUD@CSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Erika Levi, MD, MPH, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-2477
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Intrauterine Devices; Cesarean Section
Keywords: Postpartum Contraception; Intrauterine Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interval IUD Placement (No Intervention): Women randomized to this arm will be scheduled for their IUD placement 4-8 weeks after their cesarean delivery
- Immediate Postplacental IUD placement (Experimental): Women randomized to this arm will receive on IUD at time of cesarean delivery, immediately after the delivery of the placenta
  Interventions: Device: Immediate Postplacental Placement of an IUD during cesarean delivery

INTERVENTIONS:
Device: Immediate Postplacental Placement of an IUD during cesarean delivery — Women randomized to this arm will have an IUD placed during their cesarean delivery, immediately after delivery of the placenta
  Arms: Immediate Postplacental IUD placement

SUMMARY:
This is a randomized controlled trial among women who deliver by cesarean at UNC Women's Hospital and desire an Intrauterine Device (IUD) for contraception postpartum. After consenting, women will be randomized to receive an IUD at time of cesarean delivery or at a postpartum visit 4-8 weeks later. After randomization, subjects will be given a choice of the Mirena® IUD or the Paragard® IUD. Data collection will occur at baseline, delivery, the 4-8 week postpartum visit, and 2 follow-up encounters at 3 and 6 months. We hypothesize that women who receive an IUD at the time of cesarean will be more likely to use an IUD 6 months later than women who plan on receiving an IUD 4-8 weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45
* Pregnant and greater than or equal to 24 weeks of estimated gestational age
* Live Pregnancy
* States a plan to use an Intrauterine Device (IUD) postpartum for contraception
* Plan for cesarean delivery
* Intend to stay in the Chapel Hill area for at least 6 months after birth
* Fluent in English or Spanish

Exclusion Criteria:

* known uterine anomalies
* allergies to any component of the IUD of their choosing
* known or suspected carcinoma of the breast
* known acute liver disease or liver tumor (benign or malignant)
* known or suspected uterine or cervical neoplasia
* active pelvic inflammatory disease
* genital bleeding of unknown etiology
* history of solid organ transplantation
* positive test for gonorrhea or chlamydia during this pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Levi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Levi EE, Stuart GS, Zerden ML, Garrett JM, Bryant AG. Intrauterine Device Placement During Cesarean Delivery and Continued Use 6 Months Postpartum: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):5-11. doi: 10.1097/AOG.0000000000000882. PMID 26241250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement
Started | 56 | 56
Had Successful IUD Placement | 34 | 53
IUD Expulsion | 1 | 4
IUD Removal | 2 | 7
IUD in Place at 6 Months Posptartum | 32 | 40
Completed | 50 | 48
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (.51) | 28 (.57) | 28 (.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22 | 26 | 48
  Black | 15 | 13 | 28
  Hispanic | 18 | 13 | 31
  Asian | 0 | 2 | 2
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: IUD Use
Description: The use of an IUD at 6 months postpartum is the primary outcome measure
Time Frame: 6 months postpartum
Measure: Number; unit: participants
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement
Number analyzed (Participants) | 50 | 48
participants | 32 | 40

2. Secondary Outcome: IUD Expulsion
Time Frame: 0-6 months postpartum
Measure: Number; unit: participants
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement
Number analyzed (Participants) | 50 | 48
participants | 1 | 4

3. Secondary Outcome: Women's Satisfaction With IUDs
Time Frame: 0-6 months postpartum
Measure: Number; unit: percentage of participants satisfied
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement
Number analyzed (Participants) | 39 | 30
percentage of participants satisfied | 92 | 100

ADVERSE EVENTS:
Arm/Group | Interval IUD Placement | Immediate Postplacental IUD Placement
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 1/56 | 0/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interval IUD Placement (N=56) | Immediate Postplacental IUD Placement (N=56)
Uterine Perforation (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Uterine Perforation with IUD placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No